CLINICAL TRIAL: NCT02465008
Title: Analgesic Efficacy of Levobupivacaine Administration in Periprosthetic Breast Augmentation With Implants
Brief Title: Analgesic Effect of Levobupivacaine in Breast Augmentation
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Not recruiting
Sponsor: General University Hospital of Valencia (Other)
Responsible Party: Principal Investigator, Severiano Marin Bertoli, PhD, General University Hospital of Valencia
Organization: ValenciaUGH (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERPRO2014_V2
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: postoperative; Patient-reported
MeSH Terms: conditions — Pain | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- levobupivaciane group (Experimental): Levobupivacaine group (L- bupivacaine 0,25% -2,5 mg/ml-) 60 ml. Total dosis in topical use 150 mg (administered irrigation 30 ml into the surgical pocket bilaterally intraoperatively).
  Interventions: Drug: Levobupivacaine
- Placebo Comparator (saline solution) (Placebo Comparator): Placebo group (saline solution) 60 ml (administered irrigation 30 ml into the surgical pocket bilaterally intraoperatively).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levobupivacaine
  Arms: levobupivaciane group
Drug: Placebo
  Arms: Placebo Comparator (saline solution)

SUMMARY:
The purpose of this study is to determine whether levobupivacaine is effective in the acute postoperative pain treatment in periprosthetic breast augmentation

DETAILED DESCRIPTION:
One of the most common plastic surgery is breast augmentation using prosthesis ( mammoplasty Surgery with cohesive silicone gel prosthesis insubpectoral plane). Remains challenging management of acute postoperative pain that allows for early discharge of patients. To this end the following objectives are proposed: evaluate the analgesic efficacy of L-Bupivacaine 0.25% vs. Placebo (saline) administered irrigation into the surgical pocket bilaterally intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Women> 18 and <= 65 years
* Mammoplasty Surgery with cohesive silicone gel prosthesis in subpectoral plane
* ASA I and II
* Informed consent signed

Exclusion Criteria:

* Rejection of the patient
* ASA III or higher
* Other conditions that warrant their inclusion as medically indicated (eg psychiatric illness).
* Allergy to NSAIDs, local anesthetics and / or morphine
* Patients treated for chronic pain
* Placement of drains for surgical needs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Patient-reported postoperative pain. evaluated by a Visual Analog Scale (VAS) at rest and movement (cough). | at 6 hours the early postoperative period (after the end of anesthesia)